CLINICAL TRIAL: NCT07280559
Title: Evaluation of AI Medical Software-assisted LDCT Interpretation in Lung Cancer Screening and Prognosis: a Randomized Controlled Trial
Brief Title: Evaluation of AI-assisted LDCT Screening in Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Far Eastern Memorial Hospital (Other); Taipei Municipal Guandu Hospital (Unknown); Da Chien General Hospital (Other); Kinmen Hospital, Ministry of Health and Welfare (Unknown); Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2025-11-002AU-3AI
Record Dates: First submitted 2025-11-26; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-assisted LDCT Interpretation (Experimental)
  Interventions: Diagnostic Test: AI-assisted Low-Dose CT Interpretation
- Standard Radiologist LDCT Interpretation (No Intervention): Participants undergo low-dose computed tomography (LDCT) lung cancer screening. Images are interpreted solely by radiologists without AI assistance.

INTERVENTIONS:
Diagnostic Test: AI-assisted Low-Dose CT Interpretation — Participants undergo low-dose computed tomography (LDCT) lung cancer screening. The images are first interpreted by AI-assisted software, which highlights suspicious nodules. Radiologists then review the AI outputs and generate the final report.
  Arms: AI-assisted LDCT Interpretation

SUMMARY:
This multicenter pragmatic randomized controlled trial evaluates whether AI-assisted interpretation of low-dose CT (LDCT) improves lung cancer screening performance compared with standard reading. Eligible participants are randomized to AI-assisted or conventional interpretation. The study assesses diagnostic accuracy, efficiency, lung cancer incidence, mortality, recurrence, and smoking cessation outcomes. Results will inform the clinical utility and potential implementation of AI-assisted LDCT in routine screening practice.

DETAILED DESCRIPTION:
Lung cancer is a leading cause of cancer-related mortality worldwide, and early detection is essential for improving survival. Low-dose computed tomography (LDCT) has been shown to reduce lung cancer mortality in high-risk populations, but image interpretation is time-consuming and may lead to overdiagnosis. Artificial intelligence (AI)-assisted diagnostic tools offer the potential to improve accuracy and efficiency in LDCT-based lung cancer screening, though challenges related to model adaptability, data heterogeneity, user trust, and regulatory compliance remain.

This multicenter pragmatic randomized controlled trial evaluates the effectiveness of AI-assisted LDCT interpretation compared with standard interpretation. Eligible participants will be randomized to an AI-assisted arm or a standard-reading arm. Outcomes include diagnostic accuracy, efficiency, lung cancer incidence, lung cancer mortality, recurrence, and smoking cessation.

The findings will provide evidence on the clinical utility of AI-assisted LDCT screening and support future implementation in routine practice and policy development.

ELIGIBILITY:
Inclusion Criteria:

1. Family History of Lung Cancer: Males aged 45-74 or females aged 40-74 with first-degree relatives (parents, siblings, or children) diagnosed with lung cancer.
2. Heavy Smoking History: Ages 50-74 with ≥20 pack-years smoking history, currently smoking or quit <15 years ago.
3. General Screening Participants: Adults aged 40 years or older attending routine health check-ups.

Exclusion Criteria:

1. Pregnant women.
2. Chest CT or other higher-radiation chest imaging within the past 12 months.
3. Individuals holding a major illness certificate for lung cancer.
4. Inability to undergo thoracic puncture or surgery.
5. Inability to hold breath or otherwise complete the scanning procedure.
6. Hemoptysis of unknown cause within the past month.
7. Chest X-ray within the past month showing suspicious lung lesions.
8. Unexplained weight loss >6 kg within the past year.
9. History of lung cancer within the past three years.
10. Presence of other severe diseases with an expected life expectancy <5 years.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1120 (Estimated)
Dates: Start 2025-12-11 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung Cancer Incidence | From baseline to 12 months, 36 months, and 60 months.
  The proportion of newly diagnosed lung cancer cases identified within the specified follow-up period among all individuals who underwent LDCT screening.
False Positive Rate | Within 6 months following LDCT screening.
  The proportion of LDCT screening results interpreted as positive that are subsequently confirmed as non-lung cancer based on further diagnostic imaging or pathological examination.

SECONDARY OUTCOMES:
Lung Cancer Mortality | From baseline to 12 months, 36 months, and 60 months.
  The proportion of participants who die from lung cancer within the specified follow-up period after undergoing LDCT screening.
Lung Cancer Recurrence Rate | From baseline to 12 months, 36 months, and 60 months.
  The proportion of patients previously diagnosed and treated for lung cancer who experience disease recurrence during the follow-up period.
All-Cause Mortality | From baseline to 12 months, 36 months, and 60 months.
  The proportion of deaths from any cause among all individuals who underwent LDCT screening during the study period.
Time to Diagnosis | At the 12-month, 36-month, and 60-month follow-up assessments after LDCT screening.
  The time interval from LDCT screening to the date of confirmed lung cancer diagnosis, reported at the 12-month, 36-month, and 60-month follow-up time points.
Time to Treatment Initiation | At the 12-month, 36-month, and 60-month follow-up assessments after lung cancer diagnosis.
  The time interval from the date of confirmed lung cancer diagnosis to the initiation of treatment, reported at the 12-month, 36-month, and 60-month follow-up time points.
Follow-up Completion Rate | Up to 12 months post-screening.
  The proportion of individuals who completed the scheduled follow-up examinations or clinical evaluations within the designated follow-up period after undergoing LDCT screening.
Smoking Cessation Rate | Assessed at 3 months, 6 months, and 12 months after baseline screening.
  The proportion of individuals who successfully quit smoking within the follow-up period after LDCT screening

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan